CLINICAL TRIAL: NCT03255265
Title: Microchimerism and cfDNA as Biomarkers for Acute Rejection After Organ Transplantation
Brief Title: Clinical Study of Microchimerism and cfDNA as Biomarkers for Acute Rejection After Organ Transplantation
Acronym: CSMCDTITAROT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fuzhou General Hospital (Other)
Collaborators: 309th Hospital of Chinese People's Liberation Army (Other); Tianjin First Central Hospital (Other); RenJi Hospital (Other); Fudan University (Other); Ruijin Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Huazhong University of Science and Technology (Other); West China Hospital (Other); Central South University (Other); The Third Xiangya Hospital of Central South University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Qianfoshan Hospital (Other); Wuxi People's Hospital (Other); Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: cf-DNA
Record Dates: First submitted 2017-02-13; First posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-04

CONDITIONS: Organ Transplant Rejection
Keywords: organ transplantation; cfDNA; microchimerism; acute rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood

GROUPS / COHORTS (2):
- Acute rejection
  Interventions: Other: no interventions
- No acute rejection
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — no interventions

SUMMARY:
Organ transplantation has become an effective therapy for patients with end-stage organ failure at present. Rejection is still the most common cause of early dysfunction after organ transplantation. A large number of experimental and clinical data are suggesting that the formation of microchimer can successfully achieve donor-specific immune tolerance after transplantation. The formation of microchimerism may be one of the long-term survival mechanisms of transplantation, and the detection of microchimerism after transplantation can effectively predict the rejection of grafts. Scientists from Stanford University in the United States continued to report in 2014 and 2015 that using a new generation of high-throughput sequencing technology (NGS) to detect the level of free DNA from donor in blood plasma of recipients after cardiac and lung transplantation. The investigators found the level of free DNA in donor significantly increased when acute or chronic rejection happens, thus it may be used as a reflection of rejection or graft injury markers.

It has been reported that microchimerization and donor free DNA levels are associated with rejection after organ transplantation, but these studies are mostly based on a small number of cases and the results of which re qualitative and can not provide a specific microchimerization rate due to limited detection techniques. Therefore, in order to clarify the role of microchimerism and the level of cell-free DNA in donor in organ transplantation tolerance, it is necessary to use a new generation of detection technology for multi-center study with large samples.

Clinical trial was used to evaluate the clinical prediction and diagnostic value of microchimerization rate and donor cfDNA for acute rejection after organ transplantation.

950 cases of organ transplantation, of which 600 cases of renal transplantation, 300 cases of liver transplantation and 50 cases of lung transplantation.8 ml peripheral blood was collected in 1 tubes with EDTA anticoagulation. The timing of the collection was as follows: Patients with routine treatment after transplantation were preformed once every one weeks for one months and then every 3 month until the one year. In case of acute rejection, the additional blood was collected once on the day of diagnosis, and once after the treatment remission. All the samples were detected for microchimerism and cfDNA.

DETAILED DESCRIPTION:
Organ transplantation has become an effective therapy for patients with end-stage organ failure at present. Since the launch of pilot voluntary organ donation after death of citizens in 2010, the voluntary organ donation has become the only legitimate source of organ transplants in 2015, and the transition from relying on the judicial channels to obtain the organs to voluntary donation of citizens has been successfully achieved in China, donation cases and the number increased year by year. At present, the annual number of organ transplantation in China has exceeded 10,000 cases, of which kidney transplantation and liver transplantation were in the lead, respectively with more than 5000 cases and 2000 cases.

Rejection is still the most common cause of early dysfunction after organ transplantation, and the mismatching of major histocompatibility antigens (MHC, human MHC, also known as HLA) of the donor and recipient is the major cause of rejection after transplantation. Therefore, the importance of matching in organ transplantation has been widely accepted. HLA typing and HLA high resolution typing are becoming more and more common. At the same time, the latest international research shows that low-resolution HLA typing in organ transplantation also can cause significant rejection, while HLA high-resolution typing, the future trend, can improve the overall survival rate. Furthermore, NGS high-throughput sequencing will push HLA high-resolution classification to a new height.

Besides HLA matching, recipients can set up specific immune tolerance to donor grafts which will significantly affect long-term survival after operation. A large number of experimental and clinical data have suggested that the microchimerism formation can successfully facilitate donor-specific immune tolerance after transplantation. Chimera refers to the condition of the cells from the donor and from the recipient coexist and move to each other as that the donor cells exist in the recipient body after receiving the allograft or xenograft transplantation and the recipient cells exist in the graft as well. Among them, microchimera refers to the low levels of donor cells (usually less than 0.01%) in the peripheral blood circulation of transplant recipients, which is commonly seen in the patients with solid organ transplantation. The concept of microchimerism was first proposed by Thomas Starzl in the Medicine School of University of Pittsburgh in the 1990s, which pointed out that between the microchimerism and transplant immune tolerance lie a possible cause and effect relationship. The long-standing presence of microchimerism can lead to the recipient's tolerance to the donor organ. The more passer-by cells the organ has, the more cells it shifts out, making it easier to form transplantation tolerance, which explains the phenomenon of the mildest rejection after liver transplantation.

Several methods have been found to induce microchimerism, including donor-specific transfusion, donor bone marrow cell infusion, donor leukocyte infusion, spleen slice combined with organ transplantation and so on.

The formation of microchimerism is probably one of the long-term survival mechanisms of the transplanted graft, and the detection of microchimerism after transplantation can effectively predict the immune tolerance and rejection of the graft, while there is no very effective quantitation method.. In addition, the relationship between microchimerism and immunotolerance remains questionable, such as to what level of the clinical microchimerism formation that suggests stable immune tolerance, and whether it is possible to determine the withdrawal of immunosuppressive agents by the detection of microchimerism and etc., these are urgent problems remained to be solved and clarified. Based on the Insertion Deletion (InDel) site combined with quantitative real-time polymerase chain reaction, the detection sensitivity can reach 0.001% to 0.01%, which can accurately quantify the microchimerism level and dynamically monitor microchimerism after the transplantation.

At the same time, scientists from Stanford University in the United States continued to report in 2014 and 2015 that using a new generation of high-throughput sequencing technology (NGS) to detect the level of donor derived cell free DNA(cf DNA) in blood plasma of recipients after cardiac and lung transplantation. The investigators found that the level of donor-derived cf DNA was significantly increased when acute or chronic rejection happens, thus it could be used as a marker to reflect rejection or graft injury.

It has been reported that microchimerization and donor-cfDNA levels are correlated with rejection after organ transplantation, but these studies are mostly based on a small number of cases and the results of which are qualitative or with low resolution value due to limited detection techniques thus can not provide a specific microchimerism rate.

Therefore, The investigators need to clarify the role of microchimerism and the level of donor -derived cf DNA during graft injury as well as rejection after transplantation using a new generation of detection technology for multi-center study with large sample size.

In this study, 950 cases of organ transplantation, of which 600 cases of renal transplantation, 300 cases of liver transplantation and 50 cases of lung transplantation will be recruited and detected. 8 ml peripheral blood will be collected in 1 tubes with EDTA anticoagulation. The time points of the collection are as follows: Patients with routine treatment after transplantation are preformed once a week for 1 month and then at 3, 6 and 12 months after transplantation. In case of acute rejection, the additional blood will be collected once on the day of diagnosis, and once after 7 days treatment remission. All the samples were detected for microchimerism and cfDNA.

ELIGIBILITY:
Inclusion Criteria:

* Single-organ transplant recipients aged above 18 years old Recipients of re-do organ transplants
* Recipients with no systemic acute or chronic infections, infectious diseases;
* Recipients with no severe systemic diseases and/or spiritual system diseases
* Recipients or families signed the consent form.

Exclusion Criteria:

* Organ transplant recipients whose donor is child (under the age of 18 years old)
* Patients wait-listed for multiple organ transplantation
* Unable or unwilling to follow up regularly

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: aged above 18 years old single organ transplant patients (first or again); Guardian or self-signed informed consent.
Sampling Method: Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-09-28 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of the donor microchimerism in recipients was conducted once a week for 1 month and then at 3, 6 and 12 months after transplantation. | 2017.4.1-2021.4.31
  Around the 8mL peripheral whole blood was collected and the DNA in hemocytes was extracted for qPCR analysis. During which 30 target genomic genes were amplified, the donor microchimerism rate was quantified by former differentiating of InDel sites between the donor and the recipient.

SECONDARY OUTCOMES:
Quantification of the donor derived cfDNA rate in recipients was conducted once a week for 1 month and then at 3, 6 and 12 months after transplantation. | 2017.4.1-2021.4.31
  Around the 8mL peripheral whole blood was collected and the plasma was separated for following next-generation-sequencing by Illumina system (USA). The genotyping of the donor and the recipient

CONTACTS AND LOCATIONS:
Locations (1):
- Fuzhou General Hospital, Xiamen Univ Fuzhou, Fujian China, Fuzhou, Fujian, China

REFERENCES:
- [Background] Adams KM, Nelson JL. Microchimerism: an investigative frontier in autoimmunity and transplantation. JAMA. 2004 Mar 3;291(9):1127-31. doi: 10.1001/jama.291.9.1127. PMID 14996783
- [Background] Akamatsu Y, Ohkohchi N, Seya K, Satomi S. Analysis of bilirubin fraction in the bile for early diagnosis of acute rejection in living related liver transplantation. Tohoku J Exp Med. 1997 Jan;181(1):145-54. doi: 10.1620/tjem.181.145. PMID 9149349
- [Background] Aljurf M, Abalkhail H, Alseraihy A, Mohamed SY, Ayas M, Alsharif F, Alzahrani H, Al-Jefri A, Aldawsari G, Al-Ahmari A, Belgaumi AF, Walter CU, El-Solh H, Rasheed W, Albitar M. Chimerism Analysis of Cell-Free DNA in Patients Treated with Hematopoietic Stem Cell Transplantation May Predict Early Relapse in Patients with Hematologic Malignancies. Biotechnol Res Int. 2016;2016:8589270. doi: 10.1155/2016/8589270. Epub 2016 Feb 23. PMID 27006832
- [Background] Ascher NL. Microchimerism in organ transplantation. Liver Transpl Surg. 1995 Jan;1(1):43-6. doi: 10.1002/lt.500010109. No abstract available. PMID 9346540
- [Background] Avolio AW, Gozzo ML, Forni L, Agnes S, Colacicco L, Barbaresi G, Magalini SC, Castagneto M. Mitochondrial/cytoplasmic enzyme ratio for the diagnosis of acute rejection after liver transplantation: sensitivity and specificity. Transplant Proc. 1992 Dec;24(6):2572-3. No abstract available. PMID 1361263
- [Background] Bakr MA, Nagib AM, Donia AF. Induction immunosuppressive therapy in kidney transplantation. Exp Clin Transplant. 2014 Mar;12 Suppl 1:60-9. doi: 10.6002/ect.25liver.l58. PMID 24635795
- [Background] Bamgbola O. Metabolic consequences of modern immunosuppressive agents in solid organ transplantation. Ther Adv Endocrinol Metab. 2016 Jun;7(3):110-27. doi: 10.1177/2042018816641580. Epub 2016 Mar 30. PMID 27293540
- [Background] Beck J, Oellerich M, Schulz U, Schauerte V, Reinhard L, Fuchs U, Knabbe C, Zittermann A, Olbricht C, Gummert JF, Shipkova M, Birschmann I, Wieland E, Schutz E. Donor-Derived Cell-Free DNA Is a Novel Universal Biomarker for Allograft Rejection in Solid Organ Transplantation. Transplant Proc. 2015 Oct;47(8):2400-3. doi: 10.1016/j.transproceed.2015.08.035. PMID 26518940
- [Background] Biancofiore G, Pucci L, Cerutti E, Penno G, Pardini E, Esposito M, Bindi L, Pelati E, Romanelli A, Triscornia S, Salvadorini MP, Stratta C, Lanfranco G, Pellegrini G, Del Prato S, Salizzoni M, Mosca F, Filipponi F. Cystatin C as a marker of renal function immediately after liver transplantation. Liver Transpl. 2006 Feb;12(2):285-91. doi: 10.1002/lt.20657. PMID 16447198
- [Background] Capron A, Haufroid V, Wallemacq P. Intra-cellular immunosuppressive drugs monitoring: A step forward towards better therapeutic efficacy after organ transplantation? Pharmacol Res. 2016 Sep;111:610-618. doi: 10.1016/j.phrs.2016.07.027. Epub 2016 Jul 25. PMID 27468645
- [Background] Chen Y, Tai Q, Hong S, Kong Y, Shang Y, Liang W, Guo Z, He X. Pretransplantation soluble CD30 level as a predictor of acute rejection in kidney transplantation: a meta-analysis. Transplantation. 2012 Nov 15;94(9):911-8. doi: 10.1097/TP.0b013e31826784ad. PMID 23052636
- [Background] De Vlaminck I, Martin L, Kertesz M, Patel K, Kowarsky M, Strehl C, Cohen G, Luikart H, Neff NF, Okamoto J, Nicolls MR, Cornfield D, Weill D, Valantine H, Khush KK, Quake SR. Noninvasive monitoring of infection and rejection after lung transplantation. Proc Natl Acad Sci U S A. 2015 Oct 27;112(43):13336-41. doi: 10.1073/pnas.1517494112. Epub 2015 Oct 12. PMID 26460048
- [Background] De Vlaminck I, Valantine HA, Snyder TM, Strehl C, Cohen G, Luikart H, Neff NF, Okamoto J, Bernstein D, Weisshaar D, Quake SR, Khush KK. Circulating cell-free DNA enables noninvasive diagnosis of heart transplant rejection. Sci Transl Med. 2014 Jun 18;6(241):241ra77. doi: 10.1126/scitranslmed.3007803. PMID 24944192
- [Background] Delville M, Charreau B, Rabant M, Legendre C, Anglicheau D. Pathogenesis of non-HLA antibodies in solid organ transplantation: Where do we stand? Hum Immunol. 2016 Nov;77(11):1055-1062. doi: 10.1016/j.humimm.2016.05.021. Epub 2016 May 26. PMID 27237040
- [Background] Deschaseaux F, Delgado D, Pistoia V, Giuliani M, Morandi F, Durrbach A. HLA-G in organ transplantation: towards clinical applications. Cell Mol Life Sci. 2011 Feb;68(3):397-404. doi: 10.1007/s00018-010-0581-6. Epub 2010 Nov 20. PMID 21103908
- [Background] Dragun D, Catar R, Philippe A. Non-HLA antibodies in solid organ transplantation: recent concepts and clinical relevance. Curr Opin Organ Transplant. 2013 Aug;18(4):430-5. doi: 10.1097/MOT.0b013e3283636e55. PMID 23838648
- [Background] Dragun D, Hegner B. Non-HLA antibodies post-transplantation: clinical relevance and treatment in solid organ transplantation. Contrib Nephrol. 2009;162:129-39. doi: 10.1159/000170845. Epub 2008 Oct 31. PMID 19001820
- [Background] Duan Z, Zhang Y, Pan F, Zhang T, Zeng Z, Wang S, Li G, Shen B, Gao J. Association between CTLA4 gene polymorphisms and acute rejection of kidney transplantation: a meta-analysis. J Nephrol. 2012 Nov-Dec;25(6):996-1002. doi: 10.5301/jn.5000082. PMID 22307437
- [Background] Eigler J. [The acute rejection reaction following kidney transplantation. Diagnostic and therapeutic aspects]. Med Klin. 1978 Dec 1;73(48):1682-9. No abstract available. German. PMID 364275
- [Background] Eikmans M, van Halteren AG, van Besien K, van Rood JJ, Drabbels JJ, Claas FH. Naturally acquired microchimerism: implications for transplantation outcome and novel methodologies for detection. Chimerism. 2014;5(2):24-39. doi: 10.4161/chim.28908. PMID 24762743
- [Background] Elahimehr R, Scheinok AT, McKay DB. Hematopoietic stem cells and solid organ transplantation. Transplant Rev (Orlando). 2016 Oct;30(4):227-34. doi: 10.1016/j.trre.2016.07.005. Epub 2016 Aug 3. PMID 27553809
- [Background] Espinel CH, Mendez-Picon G, Currier C, Novello A, Helfrich GB, Lee HM. FE Na effective in early diagnosis of acute rejection after kidney transplantation. Proc Clin Dial Transplant Forum. 1979;9:256-9. No abstract available. PMID 399517
- [Background] Gambato M, Lens S, Fernandez-Carrillo C, Alfaro I, Forns X. Viral hepatitis and liver transplantation: pathogenesis, prevention and therapy of recurrent disease. Dig Dis. 2014;32(5):538-44. doi: 10.1159/000360831. Epub 2014 Jul 14. PMID 25034286
- [Background] Garcia Moreira V, Prieto Garcia B, Baltar Martin JM, Ortega Suarez F, Alvarez FV. Cell-free DNA as a noninvasive acute rejection marker in renal transplantation. Clin Chem. 2009 Nov;55(11):1958-66. doi: 10.1373/clinchem.2009.129072. Epub 2009 Sep 3. PMID 19729469
- [Background] Germani G, Rodriguez-Castro K, Russo FP, Senzolo M, Zanetto A, Ferrarese A, Burra P. Markers of acute rejection and graft acceptance in liver transplantation. World J Gastroenterol. 2015 Jan 28;21(4):1061-8. doi: 10.3748/wjg.v21.i4.1061. PMID 25632178
- [Background] Gielis EM, Ledeganck KJ, De Winter BY, Del Favero J, Bosmans JL, Claas FH, Abramowicz D, Eikmans M. Cell-Free DNA: An Upcoming Biomarker in Transplantation. Am J Transplant. 2015 Oct;15(10):2541-51. doi: 10.1111/ajt.13387. Epub 2015 Jul 16. PMID 26184824
- [Background] Gierej B, Kobryn K, Gierej P, Gornicka B. C4d in acute rejection after liver transplantation and its usefulness in differential diagnosis between acute liver rejection and hepatitis C recurrence. Ann Transplant. 2014 Aug 1;19:373-81. doi: 10.12659/AOT.890234. PMID 25082343
- [Background] Gozzo ML, Avolio AW, Colacicco L, Agnes S, Forni F, Barbaresi G, Castagneto M. Mitochondrial liver enzymes and the ratio between mitochondrial and cytoplasmic enzymes in the differential diagnosis of acute rejection after liver transplantation. Transplant Proc. 1993 Apr;25(2):1760-1. No abstract available. PMID 8097065